CLINICAL TRIAL: NCT00663975
Title: An Open-Label, Multi-Center Safety and Efficacy Study of DCI-1020 in Pediatric Cystic Fibrosis Patients With Exocrine Pancreatic Insufficiency
Brief Title: Open Label Safety Study of DCI-1020 in Pediatric Cystic Fibrosis (CF) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not being conducted
Sponsor: Digestive Care, Inc. (Industry)
Responsible Party: William Humphries, Digestive Care Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCI 07-001
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Digestive System Diseases; Pancreatic Disease; Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: cystic fibrosis; pancreatic insufficiency; pancreatic enzymes; pediatrics
MeSH Terms: conditions — Digestive System Diseases; Pancreatic Diseases; Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): DCI-1020 Capsules contain an enteric-coated buffered microspheres of pancrelipase, encapsulated in clear capsules. Capsules are equivalent to 4,000 USP units of lipase
  Interventions: Drug: DCI 1020

INTERVENTIONS:
Drug: DCI 1020 — capsules (4,000 units of lipase) will be administered with meals and snacks

SUMMARY:
Hypothesis:DCI 1020 capsules are safe and effective in treating exocrine pancreatic insufficiency in CF patients <= 2 years of age.

The results of this study are intended to be submitted to the FDA as part of the NDA package for marketing approval of PANCRECARB (DCI 1020).

DETAILED DESCRIPTION:
A large body of data supporting the safety and efficacy of PANCRECARB® (pancrelipase) Capsules is available in patients above age 2. This study is being performed to gather the data to demonstrate the safety and efficacy of DCI1020 in pediatric CF patients (≤ 2 years) with exocrine pancreatic insufficiency. This study also takes into consideration an "age appropriate" dosing form. Specifically, the enzymes will be administered orally by opening the capsules and emptying the microspheres into a small amount of applesauce as an example of a slightly acidic soft food such as jelly, jello, etc. for feeding.

The results of this study are intended to be submitted to the FDA as part of the NDA package for marketing approval of PANCRECARB® DCI 1020(pancrelipase).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≤ 2 years of age
* Confirmed diagnosis of CF based on the following criteria:
* One or more clinical features consistent with the CF phenotype, AND
* Positive sweat chloride ≥ 60 mEq/liter (by pilocarpine iontophoresis), OR
* Genotype with two identifiable mutations consistent with CF
* Adequate nutritional status
* Pancreatic insufficiency documented by spot fecal elastase-1 (FE 1) greater or equal to 100 micrograms/g stool
* Clinically stable with no evidence of an acute medical condition
* Parent/Guardian able to understand and sign a written informed consent and comply with the requirements of the study

Exclusion Criteria:

* History of fibrosing colonopathy
* History of being refractory to pancreatic enzyme replacement therapy
* Solid organ transplant
* History of intra-abdominal surgery
* A current diagnosis or a history of distal intestinal obstruction syndrome (DIOS) in the past six (6) months, or 2 or more episodes of DIOS in the past twelve (12) months
* Conditions known to increase fecal fat loss including: inflammatory bowel disease , celiac disease, Crohn's disease, tropical Sprue, Whipple's disease
* A known contraindication, sensitivity or hypersensitivity to porcine pancreatic enzymes
* Active liver disease with liver enzymes (alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT) or bilirubin ≥ 3 times the upper limit of normal
* Acute pancreatitis or acute exacerbation of chronic pancreatitis
* Antibiotic use as follows:
* Acute treatment with any systemic (oral or IV) antibiotics two (2) weeks prior to screening
* Treatment with erythromycin and unwilling to discontinue the treatment two (2) weeks prior to the screening. (azithromycin is allowed)
* Change in chronic treatment with systemic (oral and IV) antibiotics during the trial

NOTE:

Study patient may remain on a chronic regimen of systemic (oral or IV) antibiotics (with exception of erythromycin), if he/she started the antibiotics at least 2 weeks prior to study screening, was at his/her usual bowel pattern at the time of screening, and does not stop or change these antibiotics during the study.

* Receiving enteral tube feeding during the study
* Breast feeding during the study (expressed breast milk may be used, but not feeding at the breast)
* Expected inability to cooperate with or be non-adherent to required study procedures
* Use of narcotics
* Poorly controlled diabetes
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing, within 30 days of screening visit
* A medical condition which the investigator deems significant enough to interfere with the ability of the study patient to participate in the trial or interfering with assessment of effects of enzyme therapy on fat absorption

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Quantitative fecal fat content (%of fat/g of dry stool) in the spot stool samples collected over the 3 day In-home Treatment Period | 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Sipos, PhD, Study Director — DCI
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States